CLINICAL TRIAL: NCT03718377
Title: The Effects of Ultrasound-guided Serratus Plane Block in Combination With General Anesthesia on Intraoperative Opioid Consumption, Emergence Time and Hemodynamic Stability During Video-assisted Thoracoscopic Lobectomy
Brief Title: The Effects of Ultrasound-guided Serratus Plane Block During Video-assisted Thoracoscopic Lobectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kyungpook National University Hospital (Other)
Responsible Party: Principal Investigator, Saeyoung Kim, MD, PhD, Associate professor, Kyungpook National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018-06-006-002
Record Dates: First submitted 2018-10-18; First posted 2018-10-24 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Anesthesia, Conduction; Pain Management
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Serratus plane block (Experimental): The subjects were received serratus plane block in the regional-anesthesia unit out of operation room before induction of general anesthesia. And, video-assisted thoracic surgery was performed under balanced general anesthesia.
  Interventions: Procedure: Serratus plane block
- General anesthesia only (Active Comparator): Video-assisted thoracic surgery was performed under balanced general anesthesia without serratus plane block
  Interventions: Procedure: General anesthesia only

INTERVENTIONS:
Procedure: Serratus plane block — The subjects were received serratus plane block in the regional-anesthesia unit out of operation room before induction of general anesthesia. And, video-assisted thoracic surgery was performed under balanced general anesthesia.
  Arms: Serratus plane block
Procedure: General anesthesia only — Video-assisted thoracic surgery was performed under balanced general anesthesia without serratus plane block
  Arms: General anesthesia only

SUMMARY:
This study evaluates the effects of serratus plane block on intraoperative opioid consumption, emergence time and hemodynamic stability in patients undergoing video-assisted thoracic surgery.

DETAILED DESCRIPTION:
Thoracotomy is known as one of the most painful surgery. Thus, there is a development to reduce surgical stress in terms of operation technique, which is video-assisted thoracoscopic surgery. Although it has reduced postoperative pain and complications compared with thoracotomy, VATS is still quite painful operation.

Serratus plane block is a novel technique which provide analgesic effect for lateral chest wall by blocking lateral branch of intercostal nerve. It has been reported to be used for pain management including rib fracture, herpes zoster, and postoperative pain. It has become a popular analgesic modality because it is easy to perform and relatively safe. However, the effect of serratus plane block during intraoperative period has not yet been studied.

In this study, therefore, the investigators decided to assess the effect of serratus plane block on intraoperative opioid consumption, emergence time and hemodynamic stability in patients undergoing video-assisted thoracic surgery.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status classification I-III for three port video-assisted thoracic surgery lobectomy under general anesthesia

Exclusion Criteria:

* History of allergic reaction to local anesthetics, coagulopathy, local infection at the injection site, and systemic infection.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-08-28 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Intraoperative remifentanil consumption | through study completion, an average of 1 year
  Intraoperative remifentanil consumption will be checked.

SECONDARY OUTCOMES:
Emergence time | through study completion, an average of 1 year
  Emergence time is duration between the end of surgery and extubation. Emergence time will be checked.
Systolic blood pressure | through study completion, an average of 1 year
  Systolic blood pressure (mmHg) will be checked
Heart rate | through study completion, an average of 1 year
  Heart rate (beats per minute) will be checked
Dose of rescue drugs used to control blood pressure and HR | through study completion, an average of 1 year
  Dose of rescue drugs used to control blood pressure and HR will be checked

CONTACTS AND LOCATIONS:
Overall Officials: Saeyoung Kim, Principal Investigator — Kyungpook National University Hospital
Locations (1):
- Kyungpook national university hospital, Daegu, South Korea